CLINICAL TRIAL: NCT06394687
Title: A Randomized Cross-over Study of The Digestion of Protein Powders in Healthy Participants Using SIMBA and LIMBA Capsule
Brief Title: The Digestion of Protein Powders in Healthy Participants Using SIMBA and LIMBA Capsule
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nimble Science Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NIMCSF162
Record Dates: First submitted 2024-04-05; First posted 2024-05-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Amino Acid Change; Food Science; Nutrition; Digestion Rate; Microtia
Keywords: Mircobiome
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, crossover, clinical study in healthy participants comparing the effect of a single ingestion of MPC/FP vs MCI/SP protein powder formulations on small intestinal proteomic profile and gastric emptying. The study will enroll up to 20 healthy participants who will consume both MCP/FP and MCI/SP products in randomized order with a washout period in between. Randomization will occur in blocks of 4, with two participants per product.
Who Masked: Participant
Masking Description: Protein powders are identical in appearance and tase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPC/FP to MCI/SP (Active Comparator): Participants ingest the MPC/FP protein product for their first intervention period, then MCI/SP for their second intervention period.
  Interventions: Dietary Supplement: Milk Protein Concentrate; Dietary Supplement: Micellar Casein Isolate
- MCI/SP to MPC/FP (Active Comparator): Participants ingest the MCI/SP protein product for their first intervention period, then MPC/FP for their second intervention period.
  Interventions: Dietary Supplement: Milk Protein Concentrate; Dietary Supplement: Micellar Casein Isolate

INTERVENTIONS:
Dietary Supplement: Milk Protein Concentrate — Milk Protein Concentrate is a powdered dairy product made by removing most of the water from milk and contains a protein content below 90% on a dry matter basis. The product has been modified where some of the colloidal calcium phosphate component is reduced, which results in the dissociation of some of casein micelles, forming loose sub-micelle structures. This change modifies the digestion behaviour to be significantly faster.
  Other Names: Fast Protein
Dietary Supplement: Micellar Casein Isolate — Micellar casein isolate is a type of protein supplement derived from milk. It belongs to the casein family of proteins, which includes various forms such as micellar casein, casein hydrolysate, and caseinates. During digestion micellar casein coagulates with both gastric acidification and enzymatic hydrolysis by pepsin, forming large stable curds which slow gastric emptying and provide a slower absorption of amino acids over time.
  Other Names: Slow Protein

SUMMARY:
This study aims to understand how the Milk Protein Concentrate/Fast Protein (MCP/FP) investigational product (IP) compares to a control the Micellar Casein Isolate/Slow Protein (MCI/SP) product in healthy volunteers. It involves two phases where participants will try both products. The main goal is to measure the type and rate of amino acids quickly in the small intestine after consuming the protein products and how this relates to gastric emptying.

DETAILED DESCRIPTION:
This study aims to compare how MPC and MCI are digested on their journey to the colon, and how the proteins are digested once in colon. Traditional methods for sampling the small intestine have limitations, so a new capsule technology will be used for non-invasive sampling.

Understanding how protein supplements like MPC and MCI are digested is crucial for determining their effectiveness and suitability for various purposes. By comparing these two types of supplements, one can gain insights into their unique digestion profiles and how they interact with the body. Additionally, analyzing how these supplements affect blood amino acid levels and stool profiles can offer further insights into their impact on the body's metabolism and gut health.

To collect samples from the small intestine, the SIMBA Capsule (designed by Nimble Science Ltd) will be used. This device offers a simple, non-invasive, and painless alternative to obtain a sample of the small intestine, suitable for laboratory analysis. The SIMBA capsule consists of a small pill sized container within a specially coated shell and is the size of capsules available in the market for food supplements such as fish oils. When swallowed, the capsule's coated shell (which resists the acidic stomach and dissolves in the small intestine) will pass through the stomach into the small intestine. Once the shell is dissolved, the capsule can collect a fluid sample from the small intestine through the designed openings that are now exposed. Additionally, the small intestinal fluid softens a latch on a spring-loaded plunger which leads to closing the openings and sealing the sampled fluid contents within the container.

In addition, there is the LIMBA capsule, which is functionally similar to the SIMBA capsule. The only difference is that the coating of the LIMBA capsule takes longer to dissolve. This allows the LIMBA capsule to collect samples from the large intestine. The coating has no effect on the rate the capsule is expelled.

By using technology like the SIMBA/LIMBA capsule for non-invasive sampling, one can overcome the limitations of traditional methods and obtain more accurate data on the digestion of these protein supplements. This will enable one to make informed recommendations regarding their usage and potentially identify novel applications for these products in clinical and nutritional settings. Ultimately, this study aims to enhance one's understanding of protein supplement metabolism and provide evidence-based guidance for individuals seeking to optimize their dietary intake for better health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 to 55 years old at inclusion in the study, both female and male subjects.
2. Signed Informed Consent; willing & able to comply with study procedures.
3. Willing to maintain their diet and physical activity levels during the study.
4. Able to swallow a size-00 capsule (23mm length).
5. No planned change in diet or medical interventions during the study duration

Exclusion Criteria:

1. Use of regular prescription medications, including antihypertensives, anti-inflammatory drugs, corticosteroids, immunosuppressants, antidepressants, antipsychotics, anti-diabetic medications, and anti-arrhythmic agents, which in the opinion of the investigator, would adversely affect study safety or outcome.
2. Prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g., achalasia, eosinophilic esophagitis, cancer diagnosis or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.
3. History of known structural gastrointestinal abnormalities such as structures or fistulas leading to mechanical obstruction.
4. Known history abdominal radiation treatment.
5. Use of any medications in the week prior to the screening study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, GLP-1 analogues); laxative use is allowed if it is kept unchanged in the week prior to the study visit. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 hours is respected before swallowing the SIMBA/LIMBA capsules and PPI treatment is resumed only 4 hours thereafter.
6. Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
7. Any significant gastrointestinal, heart, liver, lung, kidney, blood, endocrine or nervous system disease, which in the opinion of the investigator, would adversely affect study safety or outcome.
8. Cancer diagnosis or treatment within the past year (non-melanoma skin cancers are acceptable).
9. History or diagnosis of immunological or infectious disease (hepatitis, tuberculosis, HIV, Parkinson's).
10. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration.
11. Antibiotic use (except for topical use) ≤ 12 weeks prior to screening. Potential participants may be eligible once a 12-week washout is completed.
12. Consumption of probiotic or prebiotic supplements within 1 month prior to screening. Potential participants may be eligible once a 1-month washout is completed.
13. Any prior Fecal Microbiota Transplantation.
14. Colon cleanses/bowel prep for 2 weeks
15. Pregnant or breastfeeding.
16. Planning to become pregnant.
17. Alcohol or drug abuse.
18. Milk or soy allergy
19. Lactose intolerant
20. Vegan diet

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Time to presentation of the peptides in the small intestine by SIMBA/LIMBA capsule | From 0 minute to 240 minutes after ingestion of the capsule per intervention period
  Time to presentation of IP or Control peptides to the small intestine compared within subjects, measured by proteomic analysis from SIMBA/LIMBA capsules located in the small intestine based on X-ray confirmation. eg. T-90 min IP vs T-90 min Control, T-60 min IP vs T-60 min Control, etc),

SECONDARY OUTCOMES:
Time to presentation of the peptides in the small intestine by blood analysis | From 0 minute to 240 minutes after ingestion of the protein product
  Time to presentation of IP or Control peptides to the small intestine compared within subjects, measured by total amino acid analysis from blood samples difference in small intestinal proteomic profile between IP and Control phases based on PCA plot. (Maximum difference is defined by comparing the various SIMBA/LIMBA capsules within each patient, eg. T-90 min IP vs T-90 min Control, T-60 min IP vs T-60 min Control, etc),
Determination of peptide composition | From 0 minute to 240 minutes after ingestion of the protein product per intervention period
  The composition of milk-derived peptides by proteomic analysis. Statistical and mathematical analyses be employed to characterize the peptide profiles.
Determination of proteolysis rate | From 0 minute to 240 minutes after ingestion of the protein product per intervention period
  The rate of milk-derived peptide proteolysis, gastric emptying, and nutrient absorption of IP or Control peptides. Statistical and mathematical analyses be employed to discern correlations and causative relationships among these processes.
Determination of metabolites from various samples | From 0 minute to 240 minutes after ingestion of the capsule per intervention period
  The presence of the milk-derived peptide metabolites in small intestine, feces, and blood samples, following the IP or control intervention. Method of analysis being metabolomic technology.
Characterization of microbiota composition by metagenomic analysis | From 0 minute to 240 minutes after ingestion of the capsule per intervention period
  Qualitative investigation of gut bacteria participation in the metabolism of dietary proteins, influencing the breakdown of peptides and amino acids during digestion, based on microbiome profiles compared across subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumming School of Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided